CLINICAL TRIAL: NCT00323726
Title: Trends in Incidence and Survivals for Ovarian Germ Cell Tumors: A 27-Year Population-Based Study
Status: Withdrawn | Type: Observational
Why Stopped: The study was limited to IRB Exempt chart review; not an applicable trial.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: HRRC 02-579
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Trends in Incidence and Survivals for Ovarian Germ Cell Tumors: A 27-Year Population-Based Study

DETAILED DESCRIPTION:
This is a chart review.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ovarian Germ Cell Tumors in the last 27 years.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ovarian germ cell tumors
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States